CLINICAL TRIAL: NCT03793426
Title: Post-marketing Observational Study on the Safety and Efficacy of Fibryga in Congenital Fibrinogen Deficiency
Brief Title: Safety and Efficacy of Fibryga in Congenital Fibrinogen Deficiency
Status: Terminated | Type: Observational
Why Stopped: FORMA-07 was initiated as a requirement imposed by the U.S. FDA as part of Octapharma's regulatory obligations. After approving Fibryga for treatment of acquired fibrinogen deficiency in 2024, FDA has agreed that the study may now be discontinued.
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: FORMA-07
Record Dates: First submitted 2018-12-19; First posted 2019-01-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Congenital Fibrinogen Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fibryga: Fibryga (human plasma-derived fibrinogen concentrate)
  Interventions: Biological: Fibryga

INTERVENTIONS:
Biological: Fibryga — Human plasma-derived fibrinogen concentrate

SUMMARY:
Open-label, Uncontrolled, Multicenter Observational Study on the Safety and Efficacy of Fibryga in Congenital Fibrinogen Deficiency

DETAILED DESCRIPTION:
There is a need to increase the body of data on treatment effectiveness and safety in the ultra-rare setting of congenital fibrinogen deficiency. Real-world evidence (RWE) derived from non-interventional studies can describe product utilization, demonstrate value, and facilitate benefit-risk assessments; RWE can only be fully assessed once a product is launched and used in a real-life setting.

This post-marketing, observational study is designed to collect information concerning safety, efficacy, and outcomes of Fibryga administration in routine clinical use in patients of any age with congenital afibrinogenemia or hypofibrinogenemia. Documentation of the administration of Fibryga in clinical practice for the treatment of both minor and major bleeding events (BEs) will not only enhance the knowledge on the efficacy and safety profile of Fibryga, but will also gather information that cannot be obtained in the same way in controlled clinical studies. These observational data will support the safety and efficacy data generated with Fibryga in good clinical practice (GCP) clinical studies, providing benefit for both physicians and patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with a documented diagnosis of congenital afibrinogenemia or hypofibrinogenemia expected to require on-demand in-hospital treatment for BEs with Fibryga

Exclusion Criteria:

* Bleeding disorder other than congenital fibrinogen deficiency
* Patients with acquired fibrinogen deficiency or dysfibrinogenemia
* Suspicion of an anti-fibrinogen inhibitor as indicated by previous in vivo recovery, if available, of <0.5 (mg/dL)/(mg/kg); there is currently no standard test for inhibitors
* Participation in an interventional clinical study at the time of or within 4 weeks prior to enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 25 patients with a documented diagnosis of congenital afibrinogenemia or hypofibrinogenemia are planned to be documented in this study
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
The incidence of thromboembolic adverse drug reactions (ADRs) | Day 0-28
  The incidence of thromboembolic ADRs in patients receiving Fibryga for on-demand treatment of bleeding, including major bleeding, will be documented

SECONDARY OUTCOMES:
Hemostatic efficacy of Fibryga for all bleeding events (BEs) collected in the study will be assessed by the investigator using a 4-point hemostatic efficacy scale | Within 2-24 hours following treatment of BEs
  The hemostatic efficacy of Fibryga for all BEs collected in the study will be assessed by the investigator using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'.
Dosage of Fibryga | Within 2-24 hours following treatment of BEs
  Fibryga will be individually dosed as per the locally approved package insert. Actual dosage administered will be documented
Duration of BEs | Within 2-24 hours following treatment of BEs
  Details of BE duration will be documented
Incidence of treatment-emergent adverse events (safety) | Day 0-28
  All ADRs in patients receiving Fibryga for on-demand treatment of BEs, including major BEs, will be documented

CONTACTS AND LOCATIONS:
Locations (4):
- Fakultní nemocnice Ostrava, Ostrava, Czechia
- Germany (3):
  - Gerinnungszentrum rhein-ruhr, Duisburg
  - Medizinische Klinik 2 / Institut für Transfusionsmedizin Universitätsklinikum, Frankfurt
  - Gerinnungszentrum Hochtaunus, Hamburg

IPD SHARING:
Plan to Share IPD: No